CLINICAL TRIAL: NCT05114733
Title: Individualized Vocational and Educational Support and Training for Clinical High Risk for Psychosis (InVEST)
Acronym: InVEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michelle Friedman-Yakobian, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P000689
Record Dates: First submitted 2021-10-01; First posted 2021-11-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Clinical High Risk for Psychosis
Keywords: clinical high risk for psychosis; psychosis risk syndrome; school functioning; intervention

STUDY DESIGN:
Intervention Model Description: waitlist control design
Who Masked: Outcomes Assessor
Masking Description: part 1 is open label design. Next part is RCT waiting list control design. assessors will be unaware of whether the participant was in the waiting list condition or the active condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- InVEST (Experimental): 4 month treatment condition
  Interventions: Behavioral: InVEST
- delayed invest (No Intervention): participants in delayed invest wait four months and are reassessed before taking part in the intervention

INTERVENTIONS:
Behavioral: InVEST — Individualized vocational and educational support and training -- participant works with BA level school/ work coach for four months
  Arms: InVEST

SUMMARY:
The purpose of this study is to test the efficacy of InVEST (Individualized Vocational and Educational Support and Training) for CHR-P (clinical high risk for psychosis) to address specific role functioning difficulties associated with the CHR-P phase. Our specific goals are:

1. Part 1: Preliminary open trial of InVEST (n = 8) to collect preliminary feasibility and acceptability data by providing the intervention, administering assessments, and collecting focus group and self-report feedback from open trial participants. The open trial phase will help to refine recruitment approaches and to modify the treatment manual as needed.
2. Part 2: Preliminary randomized controlled trial of InVEST vs. Delayed InVEST (DI) to explore preliminary evidence of efficacy of InVEST vs. DI (n = 30). The investigators hope to gain understanding of the feasibility of InVEST and the study's assessment procedures, and to gain a preliminary understanding of the intervention's efficacy for functioning difficulties experienced by young people at CHR-P.

DETAILED DESCRIPTION:
InVEST is a novel intervention that aims to target three clusters of mechanisms believed to be key in contributing to increasing functional impairment in CHR-P: 1) executive functioning (a cognitive mechanism), 2) increased stress sensitivity (an emotional mechanism), and 3) task initiation difficulties (a behavioral mechanism). Conceptually, these mechanisms are consistent with a CBT conceptualization of role functioning impairment, and the strategies to target each mechanism will be adapted based on existing evidence-based interventions combined with clinical expertise in CHR-P treatment. Finally, our proposed project is based on robust scientific evidence supporting the need for early intervention, targeting functional impairment and related risk factors in individuals at CHR-P.

This study will be organized in two parts:

Part 1: Manual development and a preliminary open-trial (n = 8) to guide the development and refinement of InVEST through coach experiences and study participant feedback. Participants will complete the intervention and then a post-intervention focus group, providing data on the feasibility of InVEST and to direct the development of the InVEST intervention manual.

Part 2: A small, randomized trial comparing InVEST treatment (2 groups, n = 15 each). Participants will be randomized using a delayed treatment design, with half of participants randomized into InVEST and half randomized into a 4-month Delayed InVEST (DI; 4 month wait to start). Primary outcome measures will include CHR-P symptoms; global role functioning; executive functioning; stress sensitivity; task initiation; hopelessness; and suicidality.

Overview of Intervention: InVEST for CHR-P

The investigators will develop and test the feasibility of InVEST, an educational and vocational functioning intervention designed for youth at CHR-P, ages 12-18. InVEST streamlines CBT-P principles into an intervention model geared towards vocational and educational functioning.

InVEST is delivered individually by a "coach" (BA-level clinician) who can meet with youth at the clinic, by phone/ video, or in meetings in the community to provide support for implementing goals. Generally, sessions are once a week for one hour, but can be adjusted depending on client needs. The coach communicates with and serves as a member of a coordinated specialty care team (CSC) for CHR-P and collaborates with the client's individual therapist. The coach begins by identifying the youth's individualized goals and notes any difficulties with executive functioning, task initiation, and/or frustration tolerance. The coach then works with the client and therapist to develop a plan for taking action to accomplish goals and for practicing skills for improving organization, task initiation and managing frustration.

Study Procedures

Part 1: Development Phase/Open Trial Developing InVEST Manual: The investigators will develop an InVEST manual.

Recruitment: During the first year, the investigators will recruit 8 young people meeting broad CHR-P criteria from CEDAR or CHR-P research programs. Meeting broad diagnostic CHR-P criteria will be pre-determined through routine clinic assessments. Releases of Information's will be obtained from all participants upon recruitment to allow sharing of eligibility information for study recruitment. The investigators will slightly stagger these participants into 2 overlapping cohorts, to permit modifications to the protocol.

Refine and elaborate InVEST: Refinement will be an iterative process guided by our ongoing experiences in each of the stages. Additionally, the investigators will hold a focus group with the open trial participants, to inform refining the manual, particularly the initial InVEST assessment, which aims to guide how to individualize the intervention to particular client needs. The group will hold a meeting after each stage with all investigators and consultants to review and further refine the manual, including at the end of the development phase. The investigators will make changes to increase InVEST's acceptability, efficacy, efficiency, clarity, and developmental appropriateness. The open trial will inform what protocol accommodations are needed for younger adolescents, changes in content to sessions, whether and how age affects acceptability and feasibility, and whether the intervention needs to be simplified.

Assessments: Participants and a parent/ caregiver will complete 2 assessments (screening/baseline and post-treatment). Given our small sample size, treatment feasibility and accessibility are our primary outcomes. Our secondary outcome is role functioning. The investigators will acquire demographic variables and diagnosis from CEDAR records, and the investigators will conduct assessments on the following constructs: CHR-P symptoms; executive functioning; stress sensitivity; task initiation; hopelessness; and suicidality.

Focus Group Post-intervention, all open trial participants will be invited to participate in a focus group (n=8) to provide feedback on the intervention, and to inform manual development.

Part 2: Pilot Study Phase

Aims: The goals of the pilot study are to a) collect data on the feasibility and acceptability of InVEST, b) test and refine the provider training procedures, c) refine and pilot test provider adherence and competency measures, and d) preliminary investigation of InVEST's primary outcome (role functioning) and mechanisms (executive functioning, stress sensitivity, and task initiation).

Treatments: After obtaining all relevant consent and assent forms and completing their baseline assessment, participants will be randomized to either InVEST, or to a waitlist, Delayed Invest (DI) condition. Participants in the intervention condition will receive 4 months of InVEST treatment, then complete a post-treatment assessment and then a 4-month follow-up assessment. Delayed Invest participants will participate in their usual treatment without the addition of InVEST for their 4 months. Then, they will complete the 4-month assessment and begin working with an InVEST coach for the next 4 months, followed by a post-InVEST assessment. As a result, all participants will receive 3 assessments (which will allow the study assessment clinician to remain blind to study condition). Additionally, this procedure will allow for some consideration of change during the Delayed InVEST period, and for some consideration of stability after the intervention ends, and will permit all participants to receive the intervention. InVEST will be implemented as a 4-month intervention.

Assessments: Participants and a parent/ caregiver will complete 3 assessments (intervention: screening/baseline, post-treatment, 4-month follow-up; waitlist: screening/baseline, pre-treatment, post-treatment). Given our small sample size, treatment feasibility and accessibility are our primary outcomes. Our secondary outcome is role functioning.

ELIGIBILITY:
Inclusion:

1. age 12-22,
2. can speak English,
3. meet broad CHR-P criteria based on the Structured Interview for Psychosis Risk Syndromes (SIPS),
4. shows at least mild role functioning impairment on the Global Functioning-Role scale (GF:R),
5. parent is willing to provide permission (and client is willing to assent) for invest coaches to communicate with treatment providers.

Exclusion:

1. Previously met diagnostic criteria for full psychosis on the Structured Interview for Psychosis Risk Syndromes.
2. Does not meet inclusion criteria listed above.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention- recruitment rate | baseline
  recruitment rates
Feasibility of intervention -Client Satisfaction | 4 months
  Attkisson Client Satisfaction Questionnaire is a seven item scale measuring an individual's personal experience with a service (range 7-28 with higher scores indicating greater level of satisfaction)
Feasibility of intervention- drop out | 4 months
  drop outs

SECONDARY OUTCOMES:
Role functioning | change from baseline to 4 months and baseline to 8 months
  The global functioning role scale is a 10 point scale that rates school or work functioning. The scale ranges from 1-10, with 10 indicating the highest level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Friedman-Yakoobian, PHD, Principal Investigator — Department of Psychiatry at BIDMC - a major teaching hospital of Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center/ Massachusetts Mental Health Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] West ML, Parrish EM, Friedman-Yakoobian M. Treatment outcomes for young people at clinical high risk for psychosis: Data from a specialized clinic. Early Interv Psychiatry. 2022 May;16(5):500-508. doi: 10.1111/eip.13187. Epub 2021 Jul 26. PMID 34309198
- [Result] West ML, Parrish EM, Green J, Howland C, Friedman-Yakoobian M. Individualized vocational and educational support and training for youth at clinical high risk for psychosis. Early Interv Psychiatry. 2022 May;16(5):492-499. doi: 10.1111/eip.13186. Epub 2021 Jul 26. PMID 34309187